CLINICAL TRIAL: NCT04796077
Title: Efficacy of an Educational Pop-Up Book in Preparing Children for Anesthesia: A Randomized Controlled Trial
Brief Title: Preparing Children for Anesthesia With an Educational Pop-Up Book
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Healthcare of Atlanta (Other)
Collaborators: Emory University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY00000660
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Pediatric Preoperative Anxiety, Pediatric Coping
Keywords: Preoperative education; Patient education; Preoperative anxiety; Pediatric outpatient surgery; Pediatric anesthesia

STUDY DESIGN:
Intervention Model Description: Patients were allocated via a block-randomized list to either the intervention arm (the educational pop-up book) or the control arm (standard care).
Who Masked: Outcomes Assessor
Masking Description: An observer-rated behavioral anxiety outcome was masked (raters were blinded to patient group assignments). Other measures were patient self-report (unmasked).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pop-Up Book (Experimental): Patients read an interactive pop-up book about general anesthesia induction in addition to standard consultation with an anesthesia provider.
  Interventions: Other: Pop-Up Book
- Standard Care (No Intervention): Patients received standard consultation with an anesthesia provider (standard care).

INTERVENTIONS:
Other: Pop-Up Book — Patients spent 5-10 minutes reading an illustrated pop-up book that promoted active learning about the process of general anesthesia induction.
  Arms: Pop-Up Book

SUMMARY:
The study evaluated an educational pop-up book about general anesthesia induction as an interactive, child-focused preoperative education resource for pediatric patients undergoing outpatient surgery. The study's objectives were to evaluate the book as an educational tool and to understand the book's effects on patient and caregiver perceptions of the surgical experience. The study's hypotheses were that preoperative education from the pop-up book, compared to standard care, would more effectively reduce children's fear and expected pain, facilitate more positive views of the procedure and preoperative explanations, encourage adaptive coping strategies, reduce behavioral anxiety at anesthesia induction, and increase caregiver satisfaction with the surgical experience.

ELIGIBILITY:
Inclusion criteria:

* Ages 5-12 (inclusive)
* Undergoing outpatient medical procedures under general anesthesia with inhalation induction
* English-speaking
* Able to provide electronic consent/assent (legal guardian)

Exclusion criteria:

* Patients with severe developmental disabilities
* Unable to obtain electronic consent/assent from a legal guardian

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 148 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Observer-Rated Behavioral Anxiety at Anesthesia Induction as assessed by the modified Yale Preoperative Anxiety Scale-Short Form | Baseline anxiety was rated upon initial entry into the preoperative holding area; anxiety at induction was rated while patients received inhalational induction via an anesthesia mask.
  Patients' behavioral anxiety at anesthesia induction was assessed relative to baseline using the observer-rated modified Yale Preoperative Anxiety Scale-Short Form. The scale ranges from 22.92-100; higher scores indicate greater anxiety (worse outcomes). Raters were preoperative nurses and circulating nurses blinded to group assignments.

SECONDARY OUTCOMES:
Fear of Anesthesia Induction as assessed by the Children's Fear Scale | Fear was rated after education and before premedication was administered.
  Patients self-reported their fear of anesthesia induction using the Children's Fear Scale. The scale ranges from 0-4; higher scores indicate greater fear (worse outcomes).
Expected Pain from the Anesthesia Mask and During Surgery as assessed by the Faces Pain Scale-Revised | Expected pain was rated after education and before premedication was administered.
  Patients self-reported how much pain they expected (1) from the anesthesia mask and (2) while asleep for the surgical procedure using the Faces Pain Scale-Revised. The scale ranges from 0-5; higher scores indicate greater expected pain (worse outcomes).
Expectations about the Procedure, Attitudes about Anesthesia, and Views of Preoperative Explanations as assessed by a Likert-Scale Questionnaire | The outcomes were rated after education and before premedication was administered.
  Patients self-reported their perceptions of the procedure and preoperative explanations (the pop-up book or provider consultation) using a 9-item Likert-scale questionnaire. The questionnaire was scored from 1-5; higher scores indicated more positive views (better outcomes).
Self-Reported Coping Strategies for Managing the Stress of Anesthesia Induction | Patients were interviewed after education and before premedication was administered.
  In a prospective interview, patients reported coping strategies for managing the stress of anesthesia induction. Greater frequencies of adaptive coping strategies indicated better outcomes.
Caregiver Satisfaction with the Surgical Experience as assessed by a Likert-Scale Questionnaire | The questionnaire was administered after the patient underwent anesthesia induction.
  Caregivers reported their satisfaction with the surgical experience using a 10-item Likert-scale questionnaire. The questionnaire was scored from 1-5; higher scores indicated more positive views (better outcomes).

CONTACTS AND LOCATIONS:
Overall Officials: Kara K Prickett, MD, Principal Investigator — Children's Healthcare of Atlanta; Emory University School of Medicine
Locations (1):
- Children's Healthcare of Atlanta Satellite Boulevard Outpatient Surgery Center, Duluth, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (including data dictionaries) will be made available to interested researchers, in addition to study protocols, the statistical analysis plan, and the informed consent form. The data will be made available upon publication to researchers who provide a methodologically sound proposal for use in achieving the goals of the approved proposal. Proposals should be submitted to Dr Kara Prickett [kara.prickett@emory.edu].
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become available after publication.
Access Criteria: Access will be granted to researchers who provide a methodologically sound proposal for use in achieving the goals of the approved proposal. Proposals should be submitted to Dr Kara Prickett [kara.prickett@emory.edu].

REFERENCES:
- [Background] Kain ZN, Mayes LC, Caldwell-Andrews AA, Karas DE, McClain BC. Preoperative anxiety, postoperative pain, and behavioral recovery in young children undergoing surgery. Pediatrics. 2006 Aug;118(2):651-8. doi: 10.1542/peds.2005-2920. PMID 16882820
- [Background] Kain ZN, Caldwell-Andrews AA, Maranets I, McClain B, Gaal D, Mayes LC, Feng R, Zhang H. Preoperative anxiety and emergence delirium and postoperative maladaptive behaviors. Anesth Analg. 2004 Dec;99(6):1648-1654. doi: 10.1213/01.ANE.0000136471.36680.97. PMID 15562048
- [Background] Chieng YJ, Chan WC, Klainin-Yobas P, He HG. Perioperative anxiety and postoperative pain in children and adolescents undergoing elective surgical procedures: a quantitative systematic review. J Adv Nurs. 2014 Feb;70(2):243-55. doi: 10.1111/jan.12205. Epub 2013 Jul 19. PMID 23865442
- [Background] Claar RL, Walker LS, Smith CA. The influence of appraisals in understanding children's experiences with medical procedures. J Pediatr Psychol. 2002 Oct-Nov;27(7):553-63. doi: 10.1093/jpepsy/27.7.553. PMID 12228327
- [Background] Fortier MA, Chorney JM, Rony RY, Perret-Karimi D, Rinehart JB, Camilon FS, Kain ZN. Children's desire for perioperative information. Anesth Analg. 2009 Oct;109(4):1085-90. doi: 10.1213/ane.0b013e3181b1dd48. PMID 19762736
- [Background] Kain ZN, Caldwell-Andrews AA, Mayes LC, Weinberg ME, Wang SM, MacLaren JE, Blount RL. Family-centered preparation for surgery improves perioperative outcomes in children: a randomized controlled trial. Anesthesiology. 2007 Jan;106(1):65-74. doi: 10.1097/00000542-200701000-00013. PMID 17197846
- [Background] West N, Christopher N, Stratton K, Gorges M, Brown Z. Reducing preoperative anxiety with Child Life preparation prior to intravenous induction of anesthesia: A randomized controlled trial. Paediatr Anaesth. 2020 Feb;30(2):168-180. doi: 10.1111/pan.13802. Epub 2020 Jan 8. PMID 31869478
- [Background] Dalley JS, McMurtry CM. Teddy and I Get a Check-Up: A Pilot Educational Intervention Teaching Children Coping Strategies for Managing Procedure-Related Pain and Fear. Pain Res Manag. 2016;2016:4383967. doi: 10.1155/2016/4383967. Epub 2016 Apr 7. PMID 27445612
- [Background] Hatava P, Olsson GL, Lagerkranser M. Preoperative psychological preparation for children undergoing ENT operations: a comparison of two methods. Paediatr Anaesth. 2000;10(5):477-86. doi: 10.1046/j.1460-9592.2000.00537.x. PMID 11012950
- [Background] Mahajan L, Wyllie R, Steffen R, Kay M, Kitaoka G, Dettorre J, Sarigol S, McCue K. The effects of a psychological preparation program on anxiety in children and adolescents undergoing gastrointestinal endoscopy. J Pediatr Gastroenterol Nutr. 1998 Aug;27(2):161-5. doi: 10.1097/00005176-199808000-00006. PMID 9702646
- [Background] Kain ZN, MacLaren JE, Hammell C, Novoa C, Fortier MA, Huszti H, Mayes L. Healthcare provider-child-parent communication in the preoperative surgical setting. Paediatr Anaesth. 2009 Apr;19(4):376-84. doi: 10.1111/j.1460-9592.2008.02921.x. Epub 2009 Jan 27. PMID 19187045
- [Background] Heckmann M, Beauchesne MA. Pediatric perioperative education current practices: a national survey of children's hospitals in the United States. J Perioper Pract. 2013 May;23(5):100-6. doi: 10.1177/175045891302300501. PMID 23767262
- [Background] Fortier MA, Del Rosario AM, Martin SR, Kain ZN. Perioperative anxiety in children. Paediatr Anaesth. 2010 Apr;20(4):318-22. doi: 10.1111/j.1460-9592.2010.03263.x. Epub 2010 Feb 23. PMID 20199609
- [Background] Chorney JM, Kain ZN. Behavioral analysis of children's response to induction of anesthesia. Anesth Analg. 2009 Nov;109(5):1434-40. doi: 10.1213/ane.0b013e3181b412cf. Epub 2009 Aug 27. PMID 19713262
- [Background] Fortier MA, Bunzli E, Walthall J, Olshansky E, Saadat H, Santistevan R, Mayes L, Kain ZN. Web-based tailored intervention for preparation of parents and children for outpatient surgery (WebTIPS): formative evaluation and randomized controlled trial. Anesth Analg. 2015 Apr;120(4):915-22. doi: 10.1213/ANE.0000000000000632. PMID 25790213
- [Background] Liguori S, Stacchini M, Ciofi D, Olivini N, Bisogni S, Festini F. Effectiveness of an App for Reducing Preoperative Anxiety in Children: A Randomized Clinical Trial. JAMA Pediatr. 2016 Aug 1;170(8):e160533. doi: 10.1001/jamapediatrics.2016.0533. Epub 2016 Aug 1. PMID 27294708
- [Background] Ryu JH, Park SJ, Park JW, Kim JW, Yoo HJ, Kim TW, Hong JS, Han SH. Randomized clinical trial of immersive virtual reality tour of the operating theatre in children before anaesthesia. Br J Surg. 2017 Nov;104(12):1628-1633. doi: 10.1002/bjs.10684. Epub 2017 Oct 4. PMID 28975600
- [Background] Chow CH, Van Lieshout RJ, Schmidt LA, Dobson KG, Buckley N. Systematic Review: Audiovisual Interventions for Reducing Preoperative Anxiety in Children Undergoing Elective Surgery. J Pediatr Psychol. 2016 Mar;41(2):182-203. doi: 10.1093/jpepsy/jsv094. Epub 2015 Oct 17. PMID 26476281
- [Background] Felder-Puig R, Maksys A, Noestlinger C, Gadner H, Stark H, Pfluegler A, Topf R. Using a children's book to prepare children and parents for elective ENT surgery: results of a randomized clinical trial. Int J Pediatr Otorhinolaryngol. 2003 Jan;67(1):35-41. doi: 10.1016/s0165-5876(02)00359-2. PMID 12560148
- [Background] Tunney AM, Boore J. The effectiveness of a storybook in lessening anxiety in children undergoing tonsillectomy and adenoidectomy in Northern Ireland. Issues Compr Pediatr Nurs. 2013 Dec;36(4):319-35. doi: 10.3109/01460862.2013.834398. Epub 2013 Sep 30. PMID 24079908
- [Background] Kassai B, Rabilloud M, Dantony E, Grousson S, Revol O, Malik S, Ginhoux T, Touil N, Chassard D, Pereira de Souza Neto E. Introduction of a paediatric anaesthesia comic information leaflet reduced preoperative anxiety in children. Br J Anaesth. 2016 Jul;117(1):95-102. doi: 10.1093/bja/aew154. PMID 27317708
- [Derived] Cordray H, Patel C, Prickett KK. Reducing Children's Preoperative Fear with an Educational Pop-up Book: A Randomized Controlled Trial. Otolaryngol Head Neck Surg. 2022 Aug;167(2):366-374. doi: 10.1177/01945998211053197. Epub 2021 Oct 26. PMID 34699270